CLINICAL TRIAL: NCT03271528
Title: Lacosamide Effects on Alcohol Self Administration and Craving in Heavy Drinkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-36766; 1R21AA026389-01 (NIH)
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Alcohol Use Disorder
Keywords: Lacosamide; Alcohol craving; Alcohol Urge Questionnaire; Obsessive-Compulsive Drinking Scale; Visual Analog Scale; Alcohol consumption; Alcohol use disorder
MeSH Terms: conditions — Alcoholism; Alcohol Drinking | interventions — Lacosamide

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo-controlled, crossover design trial to test the effect of lacosamide on alcohol self-administration and craving following a priming dose of alcohol.This study is a within subjects design in which each subject receives both study drug (lacosamide) and placebo during participation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double-blind. Medications are over-encapsulated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lacosamide (Experimental): Lacosamide titration was done to a target dose of 300mg. Participants took 100 mg of lacosamide once on day 1, 100 mg twice per day from day 2 through day 6 (200 mg daily total), on day 7 the lacosamide dose was increased to 150 mg twice daily (300 mg daily total), and on day 8 the participant took one dose of 150 mg.
  Interventions: Drug: Lacosamide
- Placebo oral capsule (Placebo Comparator): Participants took a placebo oral capsule once on day 1, twice per day from day 2 to day 7, and once on day 8.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Lacosamide — Lacosamide titration was done to a target dose of 300mg. Participants took 100 mg of lacosamide once on day 1, 100 mg twice per day from day 2 through day 6 (200 mg daily total), on day 7 the lacosamide dose was increased to 150 mg twice daily (300 mg daily total), and on day 8 the participant took one dose of 150 mg.
  Other Names: Vimpat
  Arms: Lacosamide
Drug: Placebo oral capsule — Participants took a placebo oral capsule once on day 1, twice per day from day 2 to day 7, and once on day 8.
  Arms: Placebo oral capsule

SUMMARY:
This is a double-blind, randomized, placebo-controlled, crossover design trial tested the effect of lacosamide on alcohol self-administration and craving following a priming dose of alcohol. The specific objective of this study was to determine whether lacosamide, a novel anticonvulsant that is FDA-approved for treating partial seizures, has effects on alcohol craving and consumption.

DETAILED DESCRIPTION:
The present proposal was intended to answer the call for accelerating drug development by exploring the potential of a novel anticonvulsant, lacosamide, as a candidate medication for the treatment of alcohol use disorder (AUD). This drug, which is approved for the treatment of seizure disorders, has unique pharmacological actions that include enhancement of slow sodium channel inactivation and inhibition of collapsin response mediator protein-2 (CRMP-2). Alcohol consumption in mice that had knockdown of CRMP-2 within the nucleus accumbens was decreased from levels seen in control animals. In rodent studies, lacosamide administration has produced reductions in 'excessive' drinking and has experimentally-induced decreased expression of the CRMP-2 protein. These findings implicate CRMP-2 as playing a role in the regulation of alcohol consumption. None of the FDA-approved AUD medications or medications commonly used off-label to treat AUD target this CRMP-2 pathway, making lacosamide a promising compound for AUD drug development. The aims of this study were to: 1) test the effects of lacosamide on alcohol self-administration and craving, 2) test the effects of 7 days of lacosamide administration on cognitive function, and 3) test the effects of lacosamide on alcohol consumption and craving during a 7-day period of exposure. The effects of 7 days of lacosamide (300mg) or placebo were evaluated in a human laboratory using an alcohol self-administration methodology. In this within-subjects crossover design, heavy drinkers (N=27) were randomized to the order of exposure (lacosamide or placebo) prior to completing two alcohol self-administration trials. Subjects received a priming drink of alcohol and had access to 8 alcoholic drinks over a 2-hour period. The investigators anticipated that subjects would consume less alcohol during an alcohol self-administration trial when receiving lacosamide compared to when they are receiving placebo. Significant lacosamide-induced reductions in the quantity of alcohol self-administered are considered to be an indication that this drug may have value as an AUD medication. This study may provide a rationale for phase II clinical studies testing lacosamide with a treatment-seeking AUD population. These results should also help to spur further pre-clinical investigation into the role play by CRMP-2 in regulating both alcohol consumption and alcohol seeking behaviors.

ELIGIBILITY:
Subject Inclusion Criteria

1. 21-55 years of age
2. Can provide proof of age with state-issued or federal picture ID
3. Exceeds safe weekly drinking limits (≥14 drinks for women or ≥21 drinks for men per week)
4. Reports at least an average of one episode per week of binge drinking (>3 for women, >4 for men) in the four weeks prior to baseline screening
5. Meets DSM-5 criteria for mild alcohol use disorder or greater severity.
6. Has a smartphone to complete some of the study assessments.

Subject Exclusion Criteria

1. Currently seeking treatment for alcohol problems
2. Clinical Institute Withdrawal Assessment at >10
3. DSM-5 diagnosis of current major depression, bipolar disorder, schizophrenia, bulimia/anorexia, dementia, or a substance use disorder other than alcohol, nicotine, marijuana or caffeine
4. If female, pregnant, nursing, or have plans to become pregnant
5. If female, does not agree to use an accepted form of birth control
6. Is currently using medications for which alcohol is a contraindication
7. Has a medical or mental health condition for which further alcohol exposure at the planned dose range would be contraindicated.
8. Current risk of suicidality (MINI suicidality score greater than 8 (low risk) or Yes to the ideation question #4 of the C-SSRS)
9. Has a history of myocardial infarction, congestive heart failure, has a risk for the development of heart block, or are taking medications that can decrease conduction through the atrial ventricular node.
10. Has previous exposure to lacosamide
11. Has received any form of counseling, self-help, pharmacotherapy, or other intervention to treat AUD in the past 90 days.
12. Is unwilling to suspend use of multivitamins that contain riboflavin during study participation
13. Has urine toxicology results positive for cocaine, opioids, amphetamines, buprenorphine, methadone, or methamphetamines
14. Liver function values AST or ALT are twice the normal limit
15. GFR <80 mL/min
16. Unable to comfortably abstain from nicotine for a period of 8 hours.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Devine, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Boston University Psychiatry Research Center, Clinical Studies Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 66 subjects were consented but 39 dropped out prior to randomization in the study (ineligible after screening or lost to follow-up). A total of 27 subjects were randomized.
Groups:
- Lacosamide Then Placebo: This is a within subjects design study in which each subject receives both study drug and placebo. Subjects in this group received 7 days of lacosamide before the first alcohol self-administration trial and 7 days of placebo before the second alcohol self-administration trial.
- Placebo Then Lacosamide: This is a within subjects design study in which each subject receives both study drug and placebo. Subjects in this group received 7 days of placebo before the first alcohol self-administration trial and 7 days of lacosamide before the second alcohol self-administration trial.
Period: Medication Dispense/Exposure Period 1
Arm/Group | Lacosamide Then Placebo | Placebo Then Lacosamide
Started | 13 | 14
Completed | 11 | 12
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Participation discontinued due to COVID-19 research pause | 0 | 1
Period: Alcohol Trial 1, Washout Period 1
Arm/Group | Lacosamide Then Placebo | Placebo Then Lacosamide
Started | 11 | 12
Completed | 9 | 11
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Failed urine drug screen at time of Alcohol Trial 1 | 1 | 0
Period: Medication Dispense/Exposure Period 2
Arm/Group | Lacosamide Then Placebo | Placebo Then Lacosamide
Started | 9 | 11
Completed | 8 | 11
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Alcohol Self-Administration Trial 2
Arm/Group | Lacosamide Then Placebo | Placebo Then Lacosamide
Started | 8 | 11
Completed | 8 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 66 subjects were consented, 27 subjects were randomized, and 19 subjects completed the study. Three subjects that completed the study were omitted from statistical analysis due to not consuming any alcohol during either alcohol self-administration session.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide Then Placebo | Placebo Then Lacosamide | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.4) | 37.8 (8.2) | 36.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 8 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 3 | 1 | 4
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption in Alcohol Self-Administration Trials
Description: Alcohol consumption will be measured by using a graduated cylinder to determine the amount of alcohol given to the subject that was consumed. This outcome will be measured as standard drink units. A standard drink contains approximately 0.6 fluid ounces of pure alcohol.
Time Frame: 2 hours
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Standard Drink Units (SDU)
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
Standard Drink Units (SDU) | 3.02 (3.00) | 2.35 (2.31)

2. Secondary Outcome: Verbal Fluency: Controlled Word Association (COWAT)
Description: The Controlled Word Association (COWAT) is a verbal fluency test that measures the spontaneous production of words beginning with some designated letter. The participant is asked to name words beginning with a given letter, excluding proper nouns, for one minute and this procedure is repeated three times with a different letter each time. A different set of letters was used in each of the two alcohol self-administration trials: C-F-L and P-R-W. The examiner writes down the words provided by the participant on a piece of paper. This test is scored by counting the number of words generated by the subject for each letter, then adding the scores for each of the three letters to calculate a total test score. The lowest possible score is 0 and there is no upper limit to the score range. A higher score is indicative of better outcomes (I.e. better verbal fluency).
Time Frame: 3 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 38.19 (8.26) | 42.25 (9.75)

3. Secondary Outcome: Cognitive Function: Spatial Span Forward
Description: The Wechsler Memory Scale (WMS-III) Spatial Span test will be used to assess subjects' working memory. Subjects will be shown a sequence of block tapping and asked to repeat back an increasing number of tapped blocks in the same order. Each of the 16 items on this test is scored 0 (incorrect answer) or 1 (correct answer). The total score is calculated by adding the scores for each of the 16 items. The total score range is 0-16. Higher scores are indicative of higher levels of working memory (better outcome) and lower scores are indicative of lesser working memory function (worse outcome).
Time Frame: 10 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: correct items
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
correct items | 8.44 (2.53) | 7.75 (3.70)

4. Secondary Outcome: Cognitive Function: Spatial Span Backward
Description: The Wechsler Memory Scale (WMS-III) Spatial Span test will be used to assess subjects' working memory. Subjects will be shown a sequence of block tapping and asked to repeat back an increasing number of tapped blocks in the opposite order. Each of the 16 items on this test is scored 0 (incorrect answer) or 1 (correct answer). The total score is calculated by adding the scores for each of the 16 items. The total score range is 0-16. Higher scores are indicative of higher levels of working memory (better outcome) and lower scores are indicative of lesser working memory function (worse outcome).
Time Frame: 10 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 7.19 (2.49) | 7.62 (3.14)

5. Secondary Outcome: Cognitive Function: Digit Span Forward
Description: The Wechsler Adult Intelligence Scale (WAIS-IV) Digit Span test will be used to assess subjects' working memory. Subjects will be read and asked to repeat back an increasing number of digits in the same order. Each of the 16 items on this test is scored 0 (incorrect answer) or 1 (correct answer). The total score is calculated by adding the scores for each of the 16 items. The total score range is 0-16. Higher scores are indicative of higher levels of working memory (better outcome) and lower scores are indicative of lesser working memory function (worse outcome).
Time Frame: 10 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 10.81 (1.97) | 10.81 (2.10)

6. Secondary Outcome: Cognitive Function: Digit Span Backward
Description: The Wechsler Adult Intelligence Scale (WAIS-IV) Digit Span test will be used to assess subjects' working memory. Subjects will be read and asked to repeat back an increasing number of digits in the opposite order. Each of the 16 items on this test is scored 0 (incorrect answer) or 1 (correct answer). The total score is calculated by adding the scores for each of the 16 items. The total score range is 0-16. Higher scores are indicative of higher levels of working memory (better outcome) and lower scores are indicative of lesser working memory function (worse outcome).
Time Frame: 10 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 8.06 (1.48) | 7.62 (2.16)

7. Secondary Outcome: Cognitive Function: Digit Span Sequencing
Description: The Wechsler Adult Intelligence Scale (WAIS-IV) Digit Span test will be used to assess subjects' working memory. Subjects will be read and asked to repeat back an increasing number of digits in ascending order. Each of the 16 items on this test is scored 0 (incorrect answer) or 1 (correct answer). The total score is calculated by adding the scores for each of the 16 items. The total score range is 0-16. Higher scores are indicative of higher levels of working memory (better outcome) and lower scores are indicative of lesser working memory function (worse outcome).
Time Frame: 10 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 8.12 (2.33) | 7.62 (2.36)

8. Secondary Outcome: Alcohol Craving: Obsessive-Compulsive Drinking Scale (OCDS) Pretrial
Description: The Obsessive-Compulsive Drinking Scale (OCDS) is a quick and reliable 14-item self-rating instrument that provides a total score that measures some cognitive aspects of alcohol craving (obsessive and compulsive drinking). Each of the 14 items is scored from 0 to 4. The total score is calculated by adding the scores for each of the 14 items. The total score range is 0-56. Higher scores are indicative of more obsessive or compulsive drinking and lower scores are indicative of less obsessive or compulsive drinking.
Time Frame: 5 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
scores on a scale | 10.19 (4.79) | 12.25 (5.35)

9. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Pretrial
Description: Alcohol craving was measured by self report with the Visual Analog Scale (VAS). The VAS is a straight horizontal line with one end indicating no alcohol craving and the other end indicating intense alcohol craving. The participant marks a point on the line that matches their present amount of alcohol craving. Location of the point on the line is measured for a score range of 0-100. A lower score indicates less craving for alcohol and a higher score indicated more craving for alcohol.
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
scores on a scale | 30.25 (31.00) | 31.60 (35.65)

10. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Observation Period, Minute 10
Description: as for outcome 9
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
scores on a scale | 26.75 (20.07) | 41.87 (33.42)

11. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Observation Period, Minute 20
Description: as for outcome 9
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
scores on a scale | 35.31 (28.33) | 39.75 (34.95)

12. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Observation Period, Minute 30
Description: as for outcome 9
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 35.19 (28.85) | 37.81 (36.50)

13. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Observation Period, Minute 40
Description: as for outcome 9
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 36.87 (26.71) | 36.69 (34.50)

14. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Self-Administration Blocks 1 and 2, Minute 30
Description: as for outcome 9
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 28.00 (19.73) | 31.87 (30.66)

15. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Self-Administration Blocks 1 and 2, Minute 60
Description: as for outcome 9
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 24.94 (20.78) | 30.37 (30.38)

16. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Self-Administration Blocks 1 and 2, Minute 90
Description: as for outcome 9
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 21.62 (21.60) | 27.81 (29.52)

17. Secondary Outcome: Alcohol Craving: Visual Analog Scale (VAS) Self-Administration Blocks 1 and 2, Minute 120
Description: as for outcome 9
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 23.62 (28.78) | 29.00 (32.55)

18. Secondary Outcome: Alcohol Craving: Alcohol Urge Questionnaire (AUQ) Self-Administration Blocks 1 and 2, Minute 30
Description: The Alcohol Urge Questionnaire (AUQ) is an 8-item self report that measures the participant's urge for an alcoholic drink at the time the questionnaire is completed. Questions are in the form of a 7-point Likert scale (from strongly disagree to strongly agree) and the participant selects the extent to which they disagree or agree with the 8 statements relating to desire to drink, expectation of a desired outcome from drinking, and inability to avoid drinking if alcohol was available. Each of the 8 items is scored 1-7. The total score is calculated by adding the scores for each of the items. The total score range is 8-56. Lower scores indicate less urge for alcohol and higher scores indicate more urge for alcohol.
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 24.00 (7.54) | 23.94 (8.65)

19. Secondary Outcome: Alcohol Craving: Alcohol Urge Questionnaire (AUQ) Self-Administration Blocks 1 and 2, Minute 60
Description: as for outcome 18
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 24.88 (7.49) | 26.25 (6.70)

20. Secondary Outcome: Alcohol Craving: Alcohol Urge Questionnaire (AUQ) Self-Administration Blocks 1 and 2, Minute 90
Description: as for outcome 18
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 22.94 (7.46) | 22.00 (4.98)

21. Secondary Outcome: Alcohol Craving: Alcohol Urge Questionnaire (AUQ) Self-Administration Blocks 1 and 2, Minute 120
Description: as for outcome 18
Time Frame: 1 minute
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lacosamide | Placebo Oral Capsule
Number analyzed (Participants) | 16 | 16
score on a scale | 24.94 (9.45) | 25.44 (8.34)

ADVERSE EVENTS:
Time Frame: Up to 44 days
Description: The primary risks of this study were risks related to taking study medication, loss of confidentiality, discomfort with study procedures, overconsumption of alcohol, and interference with efforts for recovery from alcohol use disorder. These risks were adequately minimized by study design and adherence to the study protocol.
Groups:
- Lacosamide: Subjects received 7 days of lacosamide before the alcohol self-administration trial.
- Placebo: Subjects received 7 days of placebo before the alcohol self-administration trial.
Arm/Group | Lacosamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 7/16 | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lacosamide (N=16) | Placebo (N=16)
Bright yellow urine (Renal and urinary disorders) | 2 | 3
Drowsiness (General disorders) | 1 | 1
Dry mouth (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Indigestion (Gastrointestinal disorders) | 1 | 2 — General indigestion and upset stomach, bloating, gassiness
Mosquito bites (Skin and subcutaneous tissue disorders) | 1 | 0
Unpleasant taste in mouth (General disorders) | 0 | 1
Mental foginess (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated early at the discretion of the Principal Investigator due to COVID-19 restrictions on human subject research recruitment, leading to a smaller number of subjects analyzed than planned. At the time of termination, 19 subjects had completed the study compared to the target sample size of 28. Three subjects that completed the study were omitted from statistical analysis due to not consuming any alcohol during either alcohol self-administration session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT03271528/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT03271528/ICF_001.pdf